CLINICAL TRIAL: NCT03442374
Title: Lumbar Spine Muscle Degeneration Inhibits Rehabilitation-Induced Muscle
Brief Title: Lumbar Spine Muscle Degeneration Inhibits Rehabilitation-Induced Muscle Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Balgrist University Hospital (Other); Spine Institute of San Diego (Spine Zone) (Unknown)
Responsible Party: Principal Investigator, Samuel R. Ward, Professor and Vice Chair of Research, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HD088437
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Disc Degeneration; Low Back Pain
Keywords: Multifidus; Muscle; Degeneration; Lumbar Spine; Disc
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Stratified by fatty infiltration severity (n=20/group x 2 groups + non exercise controls n=20)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): A single bout of moderate intensity lumbar extensor muscle exercise.
  Interventions: Other: Exercise
- Non-exercise (No Intervention): No exercise intervention.

INTERVENTIONS:
Other: Exercise — The exercise protocol consists of 1 set of 20 repetitions (range 15-25 reps) at a rate of 5 seconds/repetitions with a starting weight of 60-80% of their computerized strength score. Patients will be instructed to target an exertion level of 7/10 on the Borg Rate of Perceived Exertion (RPE) scale within their available passive ROM range into flexion-extension
  Arms: Exercise

SUMMARY:
Low back pain (LBP) is a complex condition that affects 65-85% of the population, and is the leading musculoskeletal condition contributing to disability in the United States. Disc herniation is the most common injury and 75% of individuals undergoing surgical and rehabilitative interventions for this condition experience suboptimal or poor outcomes. These patients demonstrate disability and deficits in functional capacity, including strength and endurance of the lumbar musculature. Muscle-specific changes in individuals with LBP include altered muscle volume, fatty infiltration and fibrosis, and fiber area and type. Importantly, these changes are insensitive to rehabilitation in patients with continued chronic or recurrent symptoms. While normal disuse-related atrophy in the presence of LBP is expected, more severe or chronic pathology, such as inflammation and fiber damage, may be inducing irreversible fiber degeneration and fatty/fibrotic tissue changes that impair muscle function and recovery. While the structural and adaptive capacities of healthy muscle are well understood, muscle recovery in the presence of pathology is less clear. To address this gap in knowledge, the purpose of this project is to compare structural, physiological, and adaptive responses of muscle in the presence of acute and chronic lumbar spine pathology. The central hypothesis is that chronic injury results in a state of muscle inflammation, atrophy, fibrosis, and muscle degeneration that is not responsive to exercise. The Investigators will identify which patients respond to exercise by examining muscle hypertrophic, fibrotic, inflammatory, and adipogenic gene expression profiles. Patients will be followed for six months post-operatively to measure muscle recovery and strength.

DETAILED DESCRIPTION:
AIM: To determine the effect of exercise on induction of muscle hypertrophic, fibrotic, inflammatory, and adipogenic pathways in patients with mild versus severe fatty infiltration of the multifidus muscle. Rationale. The objectives of this aim are to 1) measure molecular responses of muscle to a well-defined bout of pre-operative exercise, and 2) to determine if baseline morphological or exercise-induced molecular responses predict muscle structural recovery and functional gains up to 6 months post-operatively.

Design. This will be a longitudinal study of 40 patients with mild (< 20%) versus severe (> 50%) fatty infiltration. Non-exercise controls will also be important and the investigators intend to use a portion of biopsied tissue from other experiments as additional controls. Prior to surgery, patients will undergo clinical and MRI examinations. Additionally, patients will undergo an exercise bout 6 hours pre-operatively, and then immediately undergo a short MRI imaging protocol to measure exercise-induced perfusion changes (IVIM). Six hours after the exercise bout, the investigators will collect biopsies of the multifidus during surgery to characterize the hypertrophic, fibrotic, adipogenic, and inflammatory responses. For primary analyses, patient groups will be selected on the basis of severity of muscle fatty infiltration. Group ages and genders will be matched because the investigators know that baseline and exercise-induced gene expression varies with age. Surgical procedure and manipulation of the disc intraoperatively will be documented to account for the potential for disc and other surgery-specific effects on muscle structure. Six months post-operatively, repeated measures of muscle structure will be made via MRI. At 6, 12, and 24 weeks, strength (isokinetic dynamometer) and patient-specific function (questionnaire data) will be obtained as per standard protocol.

Methods:

Physical Examination: A physical therapist with spine injury experience will conduct the clinical exam. Age, gender and body mass index (BMI), duration of symptoms, anti-inflammatory drug use, active and passive range of motion, provocative neural tension tests (measuring joint range of motion [ROM]), strength and endurance as measured on an isokinetic dynamometer (MedX Holdings Inc.), neurovascular status, Oswestry Disability Index (81), Baecke Physical Activity Questionnaire (BPA), Fear Avoidance Beliefs Questionnaire (FABQ), and Pain Catastrophizing Scale (PCS) are important measures that capture both physical and psychosocial factors known to be related to LBP and will be collected at the clinical site. This screen will be used to confirm that discogenic symptoms are isolated to levels below L4, which allows us to use vastus lateralis as an internal control muscle biopsy.

Clinical MRI: Standard axial, sagittal oblique, and coronal oblique MR images of the spine will be collected on all patients who are scheduled for surgery. To identify disc injury severity (Pfirrmann grade), muscle fatty infiltration (Kjaer grade), and to confirm injury location, T1 and T2 non-fat suppressed or contrast-enhanced axial and sagittal MR images of the spine joint will be used.

Multimodal MRI: Imaging will be performed in a single session on a state-of-the-art 3T MRI system (GE MR750). The quantity and distribution of spine muscle volume, fat volume, and connective tissue volume will be performed from supine scans using high-resolution (1mm3) 3D FSPGR, IDEAL fat-water separation, and UTE pulse sequences, respectively using a 32-channel spine array coil. IVIM will be used to quantify regional muscle activation in response to an exercise bout.

Exercise protocol: Prior to surgery, patients will be subjected to a lumbar spine exercise protocol on a MedX Lumbar extension dynamometer with a pelvic restraint system allowing for isolation of lumbar spine muscles. The exercise protocol consists of 1 set of 20 repetitions (range 15-25 reps) at a rate of 5 seconds/repetitions with a starting weight of 60-80% of their computerized strength score. Patients will be instructed to target an exertion level of 7/10 on the Borg Rate of Perceived Exertion (RPE) scale within their available passive ROM range into flexion-extension.

Diet protocol: Importantly, the patients will remain NPO (no food or water) after the exercise bout but will have a standardized diet for 24 hours prior to the exercise bout and surgery, which mitigates the effects of diet on gene expression (137, 150-152). Evening meals will be standardized (1900h: 11 kcal/kg; 60% carbohydrate [CHO], 25% fat [FAT], 15% protein [PRO]; 2200h (3 kcal/kg; 95% CHO, 2% FAT, 3% PRO) because meal composition can acutely impact gene and protein expression.

Harvesting and storage of muscle biopsy: Muscle biopsies will be harvested within 6 hours of the exercise bout at their scheduled surgery time. Subjects will be excluded from the analysis if their biopsies are not harvested within 1 hour of the prescribed time point. Biopsies will be obtained with a standard biopsy clamp at the middle and deep margins of the multifidus muscle as noted in Aim #1 and immediately placed in RNAlater (Qiagen) for subsequent qPCR analysis or frozen in liquid nitrogen for protein abundance/phosphorylation measurements.

qPCR and western blotting: Gene expression and protein abundance will be measured by, qPCR and western blotting, respectively. Briefly, real-time PCR will be performed in a Bio-Rad CFX384 using customized plates (PrimePCR, Bio-Rad). Target gene expression will be calculated relative to values from 18S ribosomal subunit, as preliminary findings demonstrate it to be more stable than glyceraldehyde-3-phosphate dehydrogenase (GAPDH; data not presented). For genes in which we find a greater than 3-fold change in expression, western blotting will be used to assess protein abundance, as previously described.

ELIGIBILITY:
Inclusion Criteria:

* Spine pathologies requiring un-instrumented surgery (i.e. laminectomy, laminoforaminotomy, or discectomy).
* Age 21-85 years of age.

Exclusion Criteria:

* History of lumbar spine surgery.
* Patients requiring placement of instrumentation as part of the surgical procedure (i.e. fusion).
* Diabetes.
* Neuromuscular diseases.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Multifidus Muscle Fatty Infiltration | 6 months
  (% fat at 6 months - % fat at baseline / % fat at baseline)

SECONDARY OUTCOMES:
Change in Oswestry Disability Index (ODI) | 6 Months
  Disability Questionnaire (10 questions, % scale is sum of 10 questions/50, higher score is worse), 6 months - baseline
Change in Fear Avoidance Beliefs Questionnaire (FABQ) | 6 months
  Fear Avoidance Behaviors (sumo 16 items, 0-64 scale, higher score is worse), 6 months- baseline
Change in Pain Catastrophizing Scale (PCS) | 6 months
  Pain behaviors questionnaire (sum of 13 items, 0-52 scale, higher score is worse), 6 months - baseline
Change in Activated Muscle Volume (%) | After exercise (within 5 minutes)
  (% muscle activation after exercise - % muscle activation at baseline / % muscle activation at baseline)
Change in Pain (VAS) | 6 months
  Visual Analog Scale (0-100 mm scale), 6 months - baseline
Change in Strength | 6 months
  MedEx dynamometer, Back Extensor Strength (Nm), 6 months - baseline
MYHC3 gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  Embryonic myosin heavy chain gene expression
MHY3 protein abundance (ug/mg) | 6 hours after a single exercise bout
  Embryonic myosin heavy chain protein abundance
MYOG gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  Myogenin gene expression
MYOG protein abundance (ug/mg) | 6 hours after a single exercise bout
  Myogenin protein abundance
PAX7 gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  PAX7 gene expression
PAX7 gene expression (ug/mg) | 6 hours after a single exercise bout
  PAX7 protein abundance
ANKRD2 gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  ANKRD2 gene expression
ANKRD2 protein abundance (ug/mg) | 6 hours after a single exercise bout
  ANKRD2 protein abundance
MTOR gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  MTOR gene expression
MTOR protein abundance (ug/mg) | 6 hours after a single exercise bout
  MTOR protein abundance
COL1A1 gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  COL1A1 gene expression
COL3A1 gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  COL3A1 gene expression
COL9A1 gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  COL9A1 gene expression
LOX gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  LOX gene expression
CTGF gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  CTGF gene expression
TGFB1 gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  TGFB1 gene expression
MMP1 gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  MMP1 gene expression
MMP3 gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  MMP3 gene expression
MMP9 gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  MMP9 gene expression
CEBPA gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  CEBPA gene expression
FABP4 gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  FABP4 gene expression
PPARG gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  PPARG gene expression
PPARD gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  PPARD gene expression
LEP gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  LEP gene expression
ADIPOQ gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  ADIPOQ gene expression
CASP1 gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  CASP1 gene expression
CASP3 gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  CASP3 gene expression
TNFa gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  TNFa gene expression
IL10 gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  IL10 gene expression
IL6 gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  IL6 gene expression
IL1B gene expression (delta CT/delta CT) | 6 hours after a single exercise bout
  IL1B gene expression
COL1A1 Protein abundance (ug/mg) | 6 hours after a single exercise bout
  COL1A1 Protein abundance
COL3A1 Protein abundance (ug/mg) | 6 hours after a single exercise bout
  COL3A1 Protein abundance
COL9A1 Protein abundance (ug/mg) | 6 hours after a single exercise bout
  COL9A1 Protein abundance
LOX Protein abundance (ug/mg) | 6 hours after a single exercise bout
  LOX Protein abundance
CTGF Protein abundance (ug/mg) | 6 hours after a single exercise bout
  CTGF Protein abundance
TGFB1 Protein abundance (ug/mg) | 6 hours after a single exercise bout
  TGFB1 Protein abundance
MMP1 Protein abundance (ug/mg) | 6 hours after a single exercise bout
  MMP1 Protein abundance
MMP3 Protein abundance (ug/mg) | 6 hours after a single exercise bout
  MMP3 Protein abundance
MMP9 Protein abundance (ug/mg) | 6 hours after a single exercise bout
  MMP9 Protein abundance
CEBPA Protein abundance (ug/mg) | 6 hours after a single exercise bout
  CEBPA Protein abundance
FABP4 Protein abundance (ug/mg) | 6 hours after a single exercise bout
  FABP4 Protein abundance
PPARG Protein abundance (ug/mg) | 6 hours after a single exercise bout
  PPARG Protein abundance
PPARD Protein abundance (ug/mg) | 6 hours after a single exercise bout
  PPARD Protein abundance
LEP Protein abundance (ug/mg) | 6 hours after a single exercise bout
  LEP Protein abundance
ADIPOQ Protein abundance (ug/mg) | 6 hours after a single exercise bout
  ADIPOQ Protein abundance
CASP1 Protein abundance (ug/mg) | 6 hours after a single exercise bout
  CASP1 Protein abundance
CASP3 Protein abundance (ug/mg) | 6 hours after a single exercise bout
  CASP3 Protein abundance
TNFa Protein abundance (ug/mg) | 6 hours after a single exercise bout
  TNFa Protein abundance
IL10 Protein abundance (ug/mg) | 6 hours after a single exercise bout
  IL10 Protein abundance
IL6 Protein abundance (ug/mg) | 6 hours after a single exercise bout
  IL6 Protein abundance
IL1B Protein abundance (ug/mg) | 6 hours after a single exercise bout
  IL1B Protein abundance
Change in Multifidus muscle volume (%) | baseline
  Multifidus muscle volume (cc), (6 months - baseline/baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/74/NCT03442374/ICF_000.pdf